CLINICAL TRIAL: NCT03308448
Title: Traumatic Optic Neuropathy Treatment Trial 2; Efficacy of Different Doses of Erythropoietin. A Multicenter, Double Blind RCT
Brief Title: Traumatic Optic Neuropathy Treatment Trial 2
Acronym: TONTT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Collaborators: Mashhad University of Medical Sciences (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUMS 96-03-124-31806
Record Dates: First submitted 2017-09-24; First posted 2017-10-12 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Optic Neuropathy
Keywords: Traumatic optic neuropathy; Erythropoietin; EPO; Eprex
MeSH Terms: conditions — Optic Nerve Injuries | interventions — Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: 3 treatment groups of patients with TON will receive different total dose of EPO.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are unaware of the dose of EPO. Outcome assessors are masked to the dose of EPO
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Intervention is Intra-Venous injection of Eprex or EPO [recombinant human erythropoietin, Pooyesh Darou Biopharmaceuticals CO., Tehran, Iran, 4000 unit/ml solution in prefilled syringe], 300 units/kg/day for three consecutive days (total:900/kg in 3 days)
  Interventions: Drug: Recombinant human erythropoietin
- Group 2 (Active Comparator): Intervention is Intra-Venous injection of Eprex or EPO [recombinant human erythropoietin, Pooyesh Darou Biopharmaceuticals CO., Tehran, Iran, 4000 unit/ml solution in prefilled syringe], 600 units/kg/day for three consecutive days (total:1800/kg in 3 days)
  Interventions: Drug: Recombinant human erythropoietin
- Group 3 (Active Comparator): Intervention is Intra-Venous injection of Eprex or EPO [recombinant human erythropoietin, Pooyesh Darou Biopharmaceuticals CO., Tehran, Iran, 4000 unit/ml solution in prefilled syringe], 600 units/kg/day for three consecutive days then repetition of the same treatment in month 1 (Total: 3600/kg in 2 set of 3-day treatment, 1 month apart)
  Interventions: Drug: Recombinant human erythropoietin

INTERVENTIONS:
Drug: Recombinant human erythropoietin — Intravenous administration of recombinant human erythropoietin (4000 u/vial) with different dosage for each group
  Other Names: EPO, Eprex

SUMMARY:
After introducing intravenous erythropoietin (EPO) as an option for treatment of patients with indirect traumatic optic neuropathy in 2011 and publishing non inferiority trial in Oct.2017), TONTT2 is aiming to find out the best dose and timing of EPO administration in this group of patients.

DETAILED DESCRIPTION:
Patients with TON will be visited. After being eligible to enter the study and obtaining informed consent, they will be randomly assigned into 3 groups of different total dose of intravenous administration of EPO to which patients and outcome assessors will be masked. They will be assessed at different follow up time periods with the last follow up of at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Having indirect traumatic optic neuropathy(with normal eye and fundus exam)
2. Trauma to treatment interval of 3 weeks and less
3. Age of 7 years and more

Exclusion Criteria:

1. Direct optic neuropathy,
2. Glaucoma,
3. Any retinopathy
4. Globe laceration
5. Age under 7
6. Hypertension,
7. Polycythemia,
8. Creatinin more than 3 mg/dl,
9. Sensitivity to EPO
10. Patients who have received any other form of treatment for their traumatic optic neuropathy

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Change in Mean LogMAR Best corrected visual acuity (BCVA) from 20/20 to no light perception (NLP) as assessed by Snellen visual acuity chart and analyzed based on mean LogMAR change. | Before treatment and on day 1,2,3, 7, 30, and 90 days after the treatment and through study completion, an average of 24 months
  Best corrected Visual acuity is measured (Snellen eye chart) and recorded as 20/20-20/25, 20/30, 20/40, 20, 50, 20/70, 20/100, 20/200 and then counting finger (CF), hand motion (HM), light perception (LP), and no light perception (NLP)

SECONDARY OUTCOMES:
Change in Mean Log Unit of Relative afferent pupillary defect (RAPD) from 0.3 to 1.8 log unit as assessed by Neutral density filter | Before treatment and on day 1,2,3, 7, 30, and 90 days after the treatment and through study completion, an average of 24 months
  RAPD will be measured based on six log unit of 0.3, 0.6, 0.9, 1.2, 1.5,and 1.8 in which the higher the number the higher the severity score of RAPD.
Change in Mean number of visible color plates in Color vision test book. It is from 14/14 to 0/14 as assessed by Ishihara 14-plate color test book | Before treatment and on day 1,2,3, 7, 30, and 90 days after the treatment and through study completion, an average of 24 months
  Using Ishihara 14-plate color vision test book, the color vision will be recorded as a fraction of 14 plates; e.g. 10/14. Patients with lower than 20/200 vision will have 0/14 since they can not read the color plates.
Number of patients with treatment related adverse effects as assessed by history taking (change in mood, vertigo, faint), examination (blood pressure) and blood tests (CBC, BUN, Cr., K, Na, PT, PTT, INR, Ca., Ph) | before treatment and on day 1, 2 and 3 after treatment.
  history taking (change in mood, vertigo, faint), examination (blood pressure) and blood tests (CBC, BUN, Cr., K, Na, PT, PTT, INR, Ca., Ph) will be performed before treatment and on day 1, 2 and 3 after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen B Kashkouli, MD, Study Chair — Iran University of Medical Sciences
Locations (3):
- Iran (3):
  - Iran University of Medical Sciences, Tehrān, Tehran Province
  - Mashhad University of Medical Sciences, Mashhad
  - Tehran University of Medical Sciences, Tehran

IPD SHARING:
Plan to Share IPD: Yes
All IPD information will be available at the end of the study after submitting for publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: It will be published in around February 2024 and will be available for 6 months
Access Criteria: It will be available for all the researchers

REFERENCES:
- [Background] Kashkouli MB, Pakdel F, Sanjari MS, Haghighi A, Nojomi M, Homaee MH, Heirati A. Erythropoietin: a novel treatment for traumatic optic neuropathy-a pilot study. Graefes Arch Clin Exp Ophthalmol. 2011 May;249(5):731-6. doi: 10.1007/s00417-010-1534-3. Epub 2010 Oct 2. PMID 20890611
- [Background] Entezari M, Esmaeili M, Yaseri M. A pilot study of the effect of intravenous erythropoetin on improvement of visual function in patients with recent indirect traumatic optic neuropathy. Graefes Arch Clin Exp Ophthalmol. 2014 Aug;252(8):1309-13. doi: 10.1007/s00417-014-2691-6. Epub 2014 Jul 2. PMID 24986593
- [Background] Kashkouli MB, Yousefi S, Nojomi M, Sanjari MS, Pakdel F, Entezari M, Etezad-Razavi M, Razeghinejad MR, Esmaeli M, Shafiee M, Bagheri M. Traumatic optic neuropathy treatment trial (TONTT): open label, phase 3, multicenter, semi-experimental trial. Graefes Arch Clin Exp Ophthalmol. 2018 Jan;256(1):209-218. doi: 10.1007/s00417-017-3816-5. Epub 2017 Oct 6. PMID 28986670
- [Derived] Abdolalizadeh P, Kashkouli MB, Ghazizadeh M, Pakdel F, Etezad Razavi M, Nojomi M, Abri Aghdam K, Sanjari MS, Karimi N, Ghahvehchian H, Soleimani M, Tabatabaei SA. Traumatic Optic Neuropathy Treatment Trial 2 (TONTT-2): evaluating the efficacy of different doses of erythropoietin - a multicentre, randomised, double-blind clinical trial. Br J Ophthalmol. 2025 Mar 20;109(4):525-532. doi: 10.1136/bjo-2024-325828. PMID 39461733